CLINICAL TRIAL: NCT02946632
Title: Effectiveness and Tolerability of Novel, Initial Triple Combination Therapy With Xigduo (Dapagliflozin Plus Metformin) and Saxagliptin vs. Conventional Stepwise add-on Therapy in Drug-naïve Patients With Type 2 Diabetes
Brief Title: Effectiveness & Tolerability of Novel, Initial Triple Combination Therapy vs Conventional Therapy in Type 2 Diabetes
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Korea University Anam Hospital (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Sin Gon Kim, Professor, Korea University Anam Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TRIPLE-AXEL-ESR
Record Dates: First submitted 2016-10-25; First posted 2016-10-27 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2016-10

CONDITIONS: Diabetes Mellitus, Type II
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Metformin; dapagliflozin; saxagliptin; glimepiride; Sitagliptin Phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Triple combination therapy group (Experimental): Xigduo (metformin 1000mg + dapagliflozin 10mg), saxagliptin 5mg once daily for 104 weeks
  Interventions: Drug: triple combination therapy
- Stepwise add-on therapy group (Active Comparator): * Participants were started on metformin 1000mg once daily after screening & assignment
  * At each visits, FPG and HbA1c are measured. Sequential add-on therapy regimen is described
  Interventions: Drug: Stepwise add-on therapy

INTERVENTIONS:
Drug: triple combination therapy — Xigduo (metformin 1000mg + dapagliflozin 10mg) saxagliptin 5mg
  Other Names: metformin 1000mg; dapagliflozin 10mg; saxagliptin 5mg
  Arms: Triple combination therapy group
Drug: Stepwise add-on therapy — metformin -> glimepirde -> sitagliptin
  Other Names: Metformin; Glimepiride; Sitagliptin
  Arms: Stepwise add-on therapy group

SUMMARY:
In this study, the investigators will assess the efficacy and tolerability of a novel, initial triple combination therapy with metformin, saxaglipitin, and dapagliflozin, compared to conventional stepwise add-on therapy in drug-naïve patients with recently onset type 2 diabetes.

DETAILED DESCRIPTION:
ADA/EASD guideline recommends sequential treatment approach starting with metformin, and adding other classes of anti-diabetic medications if target HbA1c is not achieved. However, several clinical studies clearly showed that initial dual or triple combination therapy was more favorable in terms of glycemic control.

A DPP-4 inhibitor saxagliptin increases serum level of GLP-1, and potentiates its action of increasing glucose-dependent insulin secretion and lowering glucagon secretion. A SGLT-2 inhibitor dapagliflozin lowers hyperglycemia via blocking SGLT-2 to increase glucosuria, that is, in an insulin-independent manner. Therefore, the mechanism of action of these drugs are complimentary to that of metformin, and all of these have a low risk of hypoglycemia and weight gain.

ELIGIBILITY:
Inclusion Criteria:

* Drug-naïve patients with type 2 diabetes by American Diabetes Association criteria
* HbA1c ≥ 8%, < 10.5% at screening
* Age ≥ 18 years, < 65 years
* Body mass index (BMI) ≥ 23 kg/m2, < 35 kg/m2
* Estimated GFR (eGFR) ≥ 60 ml/min/1.73m2

Exclusion Criteria:

* Uncontrolled hyperglycemia > 270 mg/dl after an overnight fast
* Diabetic ketoacidosis
* Type 1 diabetes
* Confirmed cardiovascular disease (acute coronary syndrome, stroke, or transient ischemic attack) within 3 months of screening
* Congestive heart failure (New York Heart Association functional class IV)
* severe hepatic dysfunction (serum levels of either AST, ALT, or alkaline phosphatase above 3 x upper limit of normal (ULN))
* alcohol abuse within the 3 months prior to informed consent that would interfere with trial participation or any ongoing condition leading to a decreased compliance to study procedures or study drug intake
* pregnant women, women with potential of pregnancy not using adequate contraception method as evaluated by the investigator, lactating women
* use of systemic glucocorticoid

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2016-12; Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients who met HbA1c < 6.5% without hypoglycaemia, weight gain, or discontinuation due to adverse events at 104 weeks | 104 weeks

SECONDARY OUTCOMES:
∙ Proportion of patients who met HbA1c < 6.5% without hypoglycaemia, weight gain, or discontinuation due to adverse events at 52 weeks | 52 weeks
Proportion of patients who met HbA1c < 7.0% without hypoglycaemia, weight gain, or discontinuation due to adverse events at 104 weeks | 104 weeks
Change in body HbA1c from baseline to week 104 | 104 weeks
Change in body weight from baseline to week 104 | 104 weeks
Change in systolic blood pressure from baseline to week 104 | 104 weeks
Changes in fat and lean mass from baseline to at 104 weeks | 104 weeks

OTHER OUTCOMES:
AEs/SAEs | 104 weeks
  hypoglycemia, GI trouble, urinary tract infection, genital infection, volume depletion, panreatitis, severe cutaneous events, hypersensitivity reactions)
  * Vital signs
  * Collection of clinical chemistry/haematology parameters

CONTACTS AND LOCATIONS:
Overall Officials: SinGon Kim, MD, Principal Investigator — 'Korea University Anam Hospital' in Seoul, Korea
Locations (1):
- Korea University Anam Hospital, Seoul, South Korea

REFERENCES:
- [Result] Klein R, Klein BE, Moss SE. Relation of glycemic control to diabetic microvascular complications in diabetes mellitus. Ann Intern Med. 1996 Jan 1;124(1 Pt 2):90-6. doi: 10.7326/0003-4819-124-1_part_2-199601011-00003. PMID 8554220
- [Result] Moss SE, Klein R, Klein BE, Meuer SM. The association of glycemia and cause-specific mortality in a diabetic population. Arch Intern Med. 1994 Nov 14;154(21):2473-9. PMID 7979844
- [Result] Intensive blood-glucose control with sulphonylureas or insulin compared with conventional treatment and risk of complications in patients with type 2 diabetes (UKPDS 33). UK Prospective Diabetes Study (UKPDS) Group. Lancet. 1998 Sep 12;352(9131):837-53. PMID 9742976
- [Result] Action to Control Cardiovascular Risk in Diabetes Study Group; Gerstein HC, Miller ME, Byington RP, Goff DC Jr, Bigger JT, Buse JB, Cushman WC, Genuth S, Ismail-Beigi F, Grimm RH Jr, Probstfield JL, Simons-Morton DG, Friedewald WT. Effects of intensive glucose lowering in type 2 diabetes. N Engl J Med. 2008 Jun 12;358(24):2545-59. doi: 10.1056/NEJMoa0802743. Epub 2008 Jun 6. PMID 18539917
- [Result] ADVANCE Collaborative Group; Patel A, MacMahon S, Chalmers J, Neal B, Billot L, Woodward M, Marre M, Cooper M, Glasziou P, Grobbee D, Hamet P, Harrap S, Heller S, Liu L, Mancia G, Mogensen CE, Pan C, Poulter N, Rodgers A, Williams B, Bompoint S, de Galan BE, Joshi R, Travert F. Intensive blood glucose control and vascular outcomes in patients with type 2 diabetes. N Engl J Med. 2008 Jun 12;358(24):2560-72. doi: 10.1056/NEJMoa0802987. Epub 2008 Jun 6. PMID 18539916
- [Result] Holman RR, Paul SK, Bethel MA, Matthews DR, Neil HA. 10-year follow-up of intensive glucose control in type 2 diabetes. N Engl J Med. 2008 Oct 9;359(15):1577-89. doi: 10.1056/NEJMoa0806470. Epub 2008 Sep 10. PMID 18784090
- [Result] Inzucchi SE, Bergenstal RM, Buse JB, Diamant M, Ferrannini E, Nauck M, Peters AL, Tsapas A, Wender R, Matthews DR; American Diabetes Association (ADA); European Association for the Study of Diabetes (EASD). Management of hyperglycemia in type 2 diabetes: a patient-centered approach: position statement of the American Diabetes Association (ADA) and the European Association for the Study of Diabetes (EASD). Diabetes Care. 2012 Jun;35(6):1364-79. doi: 10.2337/dc12-0413. Epub 2012 Apr 19. No abstract available. PMID 22517736
- [Result] Garber AJ, Abrahamson MJ, Barzilay JI, Blonde L, Bloomgarden ZT, Bush MA, Dagogo-Jack S, Davidson MB, Einhorn D, Garvey WT, Grunberger G, Handelsman Y, Hirsch IB, Jellinger PS, McGill JB, Mechanick JI, Rosenblit PD, Umpierrez GE, Davidson MH. American Association of Clinical Endocrinologists' comprehensive diabetes management algorithm 2013 consensus statement--executive summary. Endocr Pract. 2013 May-Jun;19(3):536-57. doi: 10.4158/EP13176.CS. No abstract available. PMID 23816937
- [Result] Defronzo RA. Banting Lecture. From the triumvirate to the ominous octet: a new paradigm for the treatment of type 2 diabetes mellitus. Diabetes. 2009 Apr;58(4):773-95. doi: 10.2337/db09-9028. No abstract available. PMID 19336687
- [Result] Abdul-Ghani MA, Puckett C, Triplitt C, Maggs D, Adams J, Cersosimo E, DeFronzo RA. Initial combination therapy with metformin, pioglitazone and exenatide is more effective than sequential add-on therapy in subjects with new-onset diabetes. Results from the Efficacy and Durability of Initial Combination Therapy for Type 2 Diabetes (EDICT): a randomized trial. Diabetes Obes Metab. 2015 Mar;17(3):268-75. doi: 10.1111/dom.12417. Epub 2015 Jan 7. PMID 25425451
- [Result] Lewin A, DeFronzo RA, Patel S, Liu D, Kaste R, Woerle HJ, Broedl UC. Initial combination of empagliflozin and linagliptin in subjects with type 2 diabetes. Diabetes Care. 2015 Mar;38(3):394-402. doi: 10.2337/dc14-2365. Epub 2015 Jan 29. PMID 25633662
- [Result] Rosenstock J, Hansen L, Zee P, Li Y, Cook W, Hirshberg B, Iqbal N. Dual add-on therapy in type 2 diabetes poorly controlled with metformin monotherapy: a randomized double-blind trial of saxagliptin plus dapagliflozin addition versus single addition of saxagliptin or dapagliflozin to metformin. Diabetes Care. 2015 Mar;38(3):376-83. doi: 10.2337/dc14-1142. Epub 2014 Oct 28. PMID 25352655
- [Result] Augeri DJ, Robl JA, Betebenner DA, Magnin DR, Khanna A, Robertson JG, Wang A, Simpkins LM, Taunk P, Huang Q, Han SP, Abboa-Offei B, Cap M, Xin L, Tao L, Tozzo E, Welzel GE, Egan DM, Marcinkeviciene J, Chang SY, Biller SA, Kirby MS, Parker RA, Hamann LG. Discovery and preclinical profile of Saxagliptin (BMS-477118): a highly potent, long-acting, orally active dipeptidyl peptidase IV inhibitor for the treatment of type 2 diabetes. J Med Chem. 2005 Jul 28;48(15):5025-37. doi: 10.1021/jm050261p. PMID 16033281
- [Result] List JF, Woo V, Morales E, Tang W, Fiedorek FT. Sodium-glucose cotransport inhibition with dapagliflozin in type 2 diabetes. Diabetes Care. 2009 Apr;32(4):650-7. doi: 10.2337/dc08-1863. Epub 2008 Dec 29. PMID 19114612
- [Derived] Kim NH, Lim S, Kwak SH, Moon MK, Moon JS, Lee YH, Cho HC, Lee J, Kim SG. Efficacy and tolerability of novel triple combination therapy in drug-naive patients with type 2 diabetes from the TRIPLE-AXEL trial: protocol for an open-label randomised controlled trial. BMJ Open. 2018 Sep 24;8(9):e022448. doi: 10.1136/bmjopen-2018-022448. PMID 30249630